CLINICAL TRIAL: NCT03138733
Title: A Randomized, Double-blind, Multi-center Study to Establish the Efficacy and Safety of Ceftobiprole Medocaril Compared to Daptomycin in the Treatment of Staphylococcus Aureus Bacteremia, Including Infective Endocarditis
Brief Title: Ceftobiprole in the Treatment of Patients With Staphylococcus Aureus Bacteremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPR-CS-009
Record Dates: First submitted 2017-04-27; First posted 2017-05-03 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: Ceftobiprole, daptomycin, Staphylococcus aureus; Bacteremia, bloodstream infection
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Sepsis | interventions — ceftobiprole medocaril; Daptomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ceftobiprole medocaril (Experimental): Ceftobiprole 500 mg (as 667 mg ceftobiprole medocaril)
  Interventions: Drug: Ceftobiprole medocaril
- Daptomycin (Active Comparator): Daptomycin 6 mg/kg (up to 10 mg/kg based on institutional standards), with or without aztreonam
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Ceftobiprole medocaril — Ceftobiprole 500 mg (as 667 mg ceftobiprole medocaril) as a 2 h infusion
  Arms: Ceftobiprole medocaril
Drug: Daptomycin — Daptomycin 6 mg/kg (up to 10 mg/kg based on institutional standards) as a 0.5 h infusion, with or without aztreonam
  Arms: Daptomycin

SUMMARY:
The purpose of this study was to compare the efficacy and safety of ceftobiprole medocaril versus a comparator in the treatment of patients with complicated Staphylococcus aureus bacteremia (SAB).

DETAILED DESCRIPTION:
Patients were randomized 1:1 to ceftobiprole or the comparator regimen. Randomization was stratified by study site, dialysis status, and prior antibacterial treatment use within 7 days before randomization.

The three phases of the study were:

1. Screening assessments of up to 72 hours prior to randomization
2. Randomization and subsequent active treatment with intravenous (i.v.) study drug (ceftobiprole or daptomycin ± aztreonam).
3. Post-treatment, comprising an end of trial (EOT) visit (within 72 hours of last study-drug administration), Day 35 (± 3 days), Day 42 (± 3 days), and a post-treatment evaluation (PTE) visit on Day 70 (± 5 days) post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Staphylococcus aureus bacteremia (SAB), based on at least one positive blood culture obtained within the 72 h prior to randomization
* At least one of the following signs or symptoms of bacteremia:

  1. fever (e.g.≥ 38 °C/100.4 °F measured orally)
  2. white blood cell count > 10,000 or < 4,000 cells/µL, or > 10% immature neutrophils (bands)
  3. tachycardia (heart rate > 90 bpm)
  4. hypotension (systolic blood pressure < 90 mmHg)
* At least one of the following:

  1. SAB in patients undergoing chronic intermittent hemodialysis or peritoneal dialysis
  2. Persistent SAB
  3. Definite native-valve right-sided infective endocarditis by Modified Duke's Criteria
  4. Other forms of complicated SAB
  5. Osteomyelitis (including vertebral, sternal, or long-bone osteomyelitis)
  6. Epidural or cerebral abscess
* Other inclusion criteria have been applied

Exclusion Criteria:

* Treatment with potentially effective (anti-staphylococcal) systemic antibacterial treatment for more than 48 h within the 7 days prior to randomization; Exception: Documented failure of bloodstream clearance
* Bloodstream or non-bloodstream concomitant infections with Gram-negative bacteria that are known to be non-susceptible to either ceftobiprole or aztreonam
* Left-sided infective endocarditis
* Prosthetic cardiac valves or valve support rings, cardiac pacemakers, automatic implantable cardioverter-defibrillator, or left-ventricular assist devices
* Community- or hospital-acquired pneumonia
* Opportunistic infections within 30 days prior to randomization, where the underlying cause of these infections is still active
* Requirement for continuous renal-replacement therapy
* Women who are pregnant or nursing
* Other exclusion criteria have been applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica
Locations (60):
- United States (5):
  - eStudy Site - Chula Vista - PPDS, Chula Vista, California
  - Triple O Medical Services Inc, West Palm Beach, Florida
  - Mercury Street Medical Group, Butte, Montana
  - eStudy Site - Las Vegas - PPDS, Las Vegas, Nevada
  - Remington Davis Inc., Columbus, Ohio
- Argentina (3):
  - Central Hospital de San Isidro Melchor Posse, Buenos Aires
  - Medical Institute Platense SA, La Plata
  - British Sanatorium SA, Rosario
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment "Eurohospital Plovdiv", Plovdiv, Intensive Care Clinic, Plovdiv
  - University Multiprofile Hospital for Active Treatment 'Kanev', Ruse, Department of General, Purulent-Septic, Pediatric and One Day Surgery, Rousse
  - Multiprofile Hospital for Active Treatment "Dr. Ivan Seliminski", Sliven, Anesthesiology and Intensive Care Department, Sliven
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Clinic of Purulent-Septic Surgery, Sofia
- De La Costa Clinic Ltd., Barranquilla, Colombia
- Georgia (7):
  - JSC Rustavi Central Hospital, Rustavi
  - LTD High Technology Medical Center University Clinic, Tbilisi
  - LTD Academician G. Chapidze Emergency Cardiology Center, Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - LTD Academician Vakhtang Bochorishvili Clinic, Tbilisi
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - LTD N 5 Clinikal Hospital, Tbilisi
- University Hospital Regensburg, Department of Infectious Diseases, Regensburg, Germany
- "LAIKO" General Hospital, 1st Department of Internal Medicine, Athens, Greece
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - The Baruch Padeh Medical Center, Poria Illit
  - Chaim Sheba Medical Center, Ramat Gan
  - Sieff Medical Center, Safed
  - Sourasky Medical Center, Tel Aviv
- Italy (4):
  - IRCCS-University Hospital San Martino-IST, Infectious Diseases Division, Genoa
  - University of Milan-Bicocca- S.Gerardo Hospital, Monza
  - Giuliano Isontina University Health Authority, Trieste
  - Central Friuli University Healthcare Company, Udine
- Mexico (2):
  - Fray Antonio Alcalde Guadalajara Civil Hospital, Guadalajara
  - Dr. Jose Eleuterio Gonzalez Monterrey University Hospital, Monterrey
- INDICASAT SMO / Santo Tomas Hospital, Investigation Department, Panama City, Panama
- Russia (8):
  - St. Joseph Belgorod Regional Clinical Hospital, Belgorod
  - Vinogradov Moscow Municipal Hospital, Department of Surgery #14, Moscow
  - N.I. Pirogov City Clinical Hospital #1, Moscow
  - Federal State Budget Institution "Central Clinical Hospital with Polyclinic" under the Presidential Executive Office of Russian Federation, Moscow
  - L.A. Vorokhobov City Clinical Hospital #67, Moscow
  - City Hospital #33, Nizhny Novgorod
  - Pyatigorsk City Clinical Hospital, Pyatigorsk
  - Regional Clinical Hospital, Yaroslavl
- Serbia (2):
  - Zvezdara University Medical Center, Clinic of Internal Diseases, Clinical Department of Nephrology and Metabolic Disorders with Dialysis "Prof. dr Vasilije Jovanovic", Belgrade
  - Clinical Center Kragujevac, Center for Anesthesia and Reanimation, Kragujevac
- South Africa (2):
  - Worthwhile Clinical Trials, Lakeview Hospital, Benoni
  - Mediclinic Victoria - Practice of R Moodley and MI Sarwan, Tongaat
- Spain (5):
  - Hospital del Mar, Department of Intensive Care, Barcelona
  - University Hospital de Elche, Infectious Diseases Unit, Elche
  - General University Hospital Gregorio Maranon, Infectious Diseases / Internal Medicine, Madrid
  - University Hospital Ramon y Cajal, Department of Infectious Diseases, Madrid
  - University Hospital Mutua de Terrassa, Unit of Infectious Diseases, Terrassa
- Turkey (Türkiye) (2):
  - Istanbul Kartal Kosuyolu Yuksek Ihtisas Training and Research Hospital, Istanbul
  - Ondokuz Mayis University School of Medicine, Department of Infectious Diseases, Samsun
- Ukraine (7):
  - Dnipropetrovsk I.I. Mechnykov Regional Clinical Hospital, Dnipro
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - V.T. Zaitsev Institute of General and Emergency Surgery, Kharkiv
  - Public Non-Profit Enterprise: O.O. Shalimov City Clinical Hospital #2 under Kharkiv City Council, Kharkiv
  - Communal Nonprofit Enterprise "Vinnytsia Regional Clinical Hospital named after N.I. Pirogov Vinnytsia Regional Council", Vinnytsia
  - City Clinical Hospital #3, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamed K, Engelhardt M, Jones ME, Saulay M, Holland TL, Seifert H, Fowler VG Jr. Ceftobiprole versus daptomycin in Staphylococcus aureus bacteremia: a novel protocol for a double-blind, Phase III trial. Future Microbiol. 2020 Jan;15(1):35-48. doi: 10.2217/fmb-2019-0332. Epub 2020 Jan 10. PMID 31918579
- [Result] Holland TL, Cosgrove SE, Doernberg SB, Jenkins TC, Turner NA, Boucher HW, Pavlov O, Titov I, Kosulnykov S, Atanasov B, Poromanski I, Makhviladze M, Anderzhanova A, Stryjewski ME, Assadi Gehr M, Engelhardt M, Hamed K, Ionescu D, Jones M, Saulay M, Smart J, Seifert H, Fowler VG Jr; ERADICATE Study Group. Ceftobiprole for Treatment of Complicated Staphylococcus aureus Bacteremia. N Engl J Med. 2023 Oct 12;389(15):1390-1401. doi: 10.1056/NEJMoa2300220. Epub 2023 Sep 27. PMID 37754204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized male or female patients aged ≥ 18 years who had complicated Staphylococcus aureus bacteremia (SAB).
  SAB, based on ≥ 1 positive blood culture obtained within 72 h prior to randomization, with signs or symptoms of bloodstream infection
Pre-assignment Details: A total of 390 patients were randomized and comprised the Intent-to-Treat (ITT) population (ceftobiprole n = 192; comparator n = 198). Three of these patients were excluded from the modified ITT (mITT) population: one patient in the ceftobiprole group who discontinued prior to receiving study treatment, and two patients in the ceftobiprole group who were determined by central laboratory results not to have a confirmed positive blood culture for Staphylococcus aureus at baseline
Groups:
- Ceftobiprole: Ceftobiprole 500 mg (as 667 mg ceftobiprole medocaril)
  Ceftobiprole: Ceftobiprole 500 mg as a 2 h infusion
- Daptomycin: Daptomycin 6 mg/kg, with or without aztreonam
  Daptomycin: Daptomycin 6 mg/kg (up to 10 mg/kg based on institutional standards) as a 0.5 h infusion, with or without aztreonam
Period: Overall Study
Arm/Group | Ceftobiprole | Daptomycin
Started (Intent-to-Treat (ITT) population) | 192 | 198
Modified ITT (mITT) (Three patients were excluded from the mITT population in the ceftobiprole group: one patient discontinued prior to receiving study treatment, and two patients were determined by central laboratory results not to have a confirmed positive blood culture for Staphylococcus aureus at baseline) | 189 | 198
Completed | 157 | 169
Not Completed | 35 | 29
Not completed — Death | 17 | 18
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Administrative or logistical reason | 1 | 0
Not completed — The patient was transferred to another hospital | 1 | 0

BASELINE CHARACTERISTICS:
Population: The mITT (Intent-to-Treat population who received any dose of study medication) and who had a blood culture positive for staphylococcus aureus represented the Baseline Analysis Population. It comprised 387 out of the 390 patients in the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftobiprole | Daptomycin | Total
Number analyzed (Participants) | 189 | 198 | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (15.18) | 56.5 (15.33) | 56.0 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 140 | 268
  Male | 61 | 58 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 29
  Not Hispanic or Latino | 174 | 182 | 356
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 5 | 9
  White | 179 | 192 | 371
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 175 | 185 | 360
  North America | 5 | 5 | 10
  Central America | 4 | 2 | 6
  South America | 3 | 4 | 7
  South Africa | 2 | 2 | 4
Aztreonam treatment at baseline [Count of Participants; unit: Participants] | 0 | 62 | 62
Most frequent baseline categories of complicated SAB (Investigator-assessed) [Count of Participants; unit: Participants]
  Skin and skin structure infection | 116 | 121 | 237
  Intra-abdominal abscess | 26 | 29 | 55
  Chronic dialysis | 24 | 25 | 49
  Septic arthritis | 22 | 19 | 41
  Persistent SAB | 16 | 16 | 32
  Osteomyelitis | 13 | 17 | 30
  Definite right-sided endocarditis | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With or Without Overall Success at the Post-treatment Evaluation (PTE) Visit
Description: Comparison of overall success rates in the mITT population
  Overall success at PTE for the mITT population was defined as all of the following criteria being met (Responder):
  1. Patient alive at Day 70 (± 5 days) post-randomization.
  2. No new metastatic foci or complications of the SAB infection.
  3. Resolution or improvement of SAB-related clinical signs and symptoms.
  4. Two negative blood cultures for S. aureus (without any subsequent positive blood culture for S. aureus)
Time Frame: PTE visit on Day 70 (± 5 days) post-randomization
Population: The mITT population comprised the subset of patients in the ITT population who received any dose of study medication, and had a blood culture positive for S. aureus at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 189 | 198
Participants
  Number of responders | 132 | 136
  Number of non-responders | 57 | 62
Statistical Analysis 1: Comparison: Ceftobiprole vs Daptomycin; The observed difference in percentage of responders at PTE (ceftobiprole group minus the daptomycin group) were determined and a two-sided 95% confidence interval (CI) for the observed difference was computed, with adjustment for actual stratum (dialysis status and prior antibacterial treatment use). Cochran-Mantel-Haenszel (CMH) weights were used for the stratum weight in the calculation of the CI; Test type: Non-Inferiority — The non-inferiority hypothesis test was a one-sided hypothesis test performed at the 2.5% level of significance. If the lower limit of the two sided 95% CI for the difference in response rates in the mITT population was greater than -15%, the non-inferiority of ceftobiprole to daptomycin therapy was to be concluded; Adjusted proportion difference = 2.0, 95% CI 2-sided [-7.1 to 11.1]

2. Secondary Outcome: Number of Patients With or Without Overall Success at the PTE Visit in the CE Population
Description: Comparison of overall success rates in the Clinical Evaluable (CE) population
  Overall success at PTE for the CE population was defined as all of the following criteria being met (Responder):
  1. Patient alive at Day 70 (± 5 days) post-randomization.
  2. No new metastatic foci or complications of the SAB infection.
  3. Resolution or improvement of SAB-related clinical signs and symptoms.
  4. Two negative blood cultures for S. aureus (without any subsequent positive blood culture for S. aureus)
Time Frame: At PTE visit on Day 70 (± 5 days) post-randomization
Population: The CE population comprised the subset of patients in the mITT population who complied with important pre-specified aspects of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 163 | 167
Participants
  Number of responders | 127 | 130
  Number of non-responders | 36 | 37
Statistical Analysis 1: Comparison: Ceftobiprole vs Daptomycin; Test type: Other; Adjusted proportion difference = 0.6, 95% CI 2-sided [-8.3 to 9.5] — The two-sided 95% CI was computed using Cochran-Mantel-Haenszel (CMH) weights method adjusted for actual stratum (dialysis status and prior antibacterial treatment use)

3. Secondary Outcome: Number of Patients With Microbiological Eradication at the PTE Visit
Description: Comparison of microbiological eradication rates in the mITT population. Microbiological eradication rate was defined as a negative blood culture for S. aureus during study treatment and another negative blood culture during the follow up period up to PTE.
Time Frame: At PTE visit on Day 70 (± 5 days) post-randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 189 | 198
Participants | 155 | 153
Statistical Analysis 1: Comparison: Ceftobiprole vs Daptomycin; Test type: Other; Adjusted proportion difference = 5.1, 95% CI 2-sided [-2.9 to 13] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: All-cause Mortality at the PTE Visit
Description: Comparison of all-cause mortality rates in the mITT population
Time Frame: At PTE visit on Day 70 (± 5 days) post-randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 189 | 198
Participants
  Patients died | 17 | 18
  Patients alive | 172 | 180
Statistical Analysis 1: Comparison: Ceftobiprole vs Daptomycin; Test type: Other; Adjusted proportion difference = -0.5, 95% CI 2-sided [-6.2 to 5.2] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Patients With or Without New Metastatic Foci or Other Complications of SAB Developed After Day 7
Description: Comparison of complication rates in the mITT population defined by number of patients with development of new metastatic foci or other complications of SAB after Day 7
Time Frame: Assessment after Day 7 post-randomization through to post-treatment evaluation (PTE) visit on Day 70 (± 5 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 189 | 198
Participants
  Patients with development of new metastatic foci or other complications of SAB after Day 7 | 11 | 11
  Patients without development of new metastatic foci or other complications of SAB after Day 7 | 178 | 187
Statistical Analysis 1: Comparison: Ceftobiprole vs Daptomycin; Test type: Other; Adjusted proportion difference = 0.1, 95% CI 2-sided [-4.6 to 4.8] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Time to Staphylococcus Aureus Bloodstream Clearance
Description: Time-to-event in the mITT Bloodstream clearance was defined as two consecutive study days with blood-culture-negative assessments for S. aureus, without any subsequent S. aureus relapse or reinfection
Time Frame: Up to 6 weeks post-randomization
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 189 | 198
Days | 4 [3 to 5] | 4 [3 to 5]

7. Secondary Outcome: Number of Patients With or Without Adverse Events (AEs)
Description: Treatment-emergent adverse events in the safety population
Time Frame: AEs were assessed from the first dose of study drug through the post-treatment evaluation (PTE) visit on Day 70 (± 5 days)
Population: The Safety population comprised all randomized patients who received any dose of study drug. Patients in the Safety population were analyzed according to the first study drug received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftobiprole | Daptomycin
Number analyzed (Participants) | 191 | 198
Participants
  Any adverse events (AEs) | 121 | 117
  Any drug-related AE | 25 | 11
  Any severe AEs | 29 | 38
  Any study drug-related severe AEs | 1 | 2
  Any serious adverse events (SAE) | 36 | 45
  Any drug-related SAEs | 2 | 4
  Any AE leading to treatment discontinuation | 18 | 18
  Study drug-related AEs leading to treatment discontinuation | 9 | 3
  Any AE leading to death | 17 | 18
  Study drug-related AEs leading to death | 0 | 0
  Any AE of special interest (AESI) | 9 | 7
  Any drug-related AESI | 5 | 4

ADVERSE EVENTS:
Time Frame: All AEs occurring from the start of first dosing up to and including the scheduled PTE visit on Day 70 (± 5 days) were collected.
Description: All AEs were defined as treatment-emergent AEs (TEAEs), i.e., occurring from the start of first dosing up to and including the scheduled PTE visit, and were considered for the analysis purpose.
Arm/Group | Ceftobiprole | Daptomycin
All-Cause Mortality (participants affected / at risk) | 17/191 | 18/198
Serious Adverse Events (participants affected / at risk) | 36/191 | 45/198
Other Adverse Events (participants affected / at risk) | 61/191 | 45/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftobiprole (N=191) | Daptomycin (N=198)
Wound healing normal (Investigations) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Intracardiac mass (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eosinophilic pneumonia acute (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 3
Candida sepsis (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 2
Laryngitis (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Purulent pericarditis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic necrosis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 4 | 8
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 3
Superinfection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemodialysis complication (Injury, poisoning and procedural complications) | 1 | 0
Kidney rupture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leg amputation (Surgical and medical procedures) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 1
Death (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 4 | 2
Pyrexia (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceftobiprole (N=191) | Daptomycin (N=198)
Blood potassium decreased (Investigations) | 17 | 5
Gamma-glutamyltransferase increased (Investigations) | 12 | 15
Anaemia (Blood and lymphatic system disorders) | 20 | 24
Diarrhoea (Gastrointestinal disorders) | 13 | 5
Nausea (Gastrointestinal disorders) | 20 | 8
Vomiting (Gastrointestinal disorders) | 16 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT03138733/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT03138733/SAP_001.pdf